CLINICAL TRIAL: NCT00901810
Title: Clinical Evaluation of Working Length Determination by Electronic Apex-Locator or Radiography on Adequacy of Final Working Length
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Shohre Ravanshad, DDS, MSD, Shiraz University of Medical Sciences - Dental School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sums316
Record Dates: First submitted 2009-05-12; First posted 2009-05-14 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Root Canal
Keywords: Length Determination; Working Length; Electronic Apex Locator; Root Canal Therapy; Endodontics
MeSH Terms: interventions — Radiography, Dental

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apex Locator (Active Comparator): Working length for cleaning and shaping of the canal is measured by Electronic Apex Locator in this group.
  Interventions: Device: Electronic Apex Locator
- Radiography (Active Comparator): Working length for cleaning and shaping of the canal is measured by Radiography in this group.
  Interventions: Device: Dental Radiography

INTERVENTIONS:
Device: Electronic Apex Locator — Electronic Apex Locator is used to find the apical foramen of the root canal. It uses a weak electrical current passed through the canal by endodontic file.
  Other Names: RootZX; Raypex
  Arms: Apex Locator
Device: Dental Radiography — Radiography is used to measure the length of root canal by putting an endodontic file in the canal and taking the radiography to measure the length.
  Other Names: pre apical Radiography
  Arms: Radiography

SUMMARY:
Accurate length determination of root canal is essential in root canal therapy. Radiography has been the conventional method for this measurement but recently several in-vitro studies have shown that new generations of Electronic Apex locators are as accurate as radiography in length determination. It is hypothesized that the latest generation of Electronic Apex locator can produce acceptable results as radiography when used for length determination.

ELIGIBILITY:
Inclusion Criteria:

* All the patients who are referred for Root Canal Therapy

Exclusion Criteria:

* Blocked Canals
* Open Apexes

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-07 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
adequacy of final working length | at the end of cleaning and shaping

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University of Medical Sciences - Dental School, Shiraz, Fars, Iran